CLINICAL TRIAL: NCT06940219
Title: Delayed Against Rapid Sequence Induction in Critically Ill Adults With Medical Diseases Undergoing Emergency Endotracheal Intubation: The DARSITUBE-study, a Monocentric Randomized Controlled Trial
Brief Title: Delayed Against Rapid Sequence Induction in Adults With Medical Diseases Undergoing Emergency Endotracheal Intubation.
Acronym: DARSITUBE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leipzig University Medical Center (Other)
Responsible Party: Principal Investigator, Anton Pelka, Principal Investigator, Leipzig University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 419/24-ek
Record Dates: First submitted 2025-04-07; First posted 2025-04-23 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Intubation in Intensive Care Units
Keywords: Intubation; Airway Management; Acute respiratory failure; Intensive Care Unit; Rapid Sequence Induction; Delayed Sequence Induction; Intubation in intensive care units
MeSH Terms: interventions — Rapid Sequence Induction and Intubation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RSI (Active Comparator): Modified Rapid Sequence Induction
  Interventions: Procedure: Modified Rapid Sequence Induction
- DSI (Experimental): Delayed Sequence Induction
  Interventions: Procedure: Delayed Sequence Induction

INTERVENTIONS:
Procedure: Delayed Sequence Induction — Delayed Sequence Induction - fractional dosing of Ketamin and Midazolam until a dissociative status is achieved. Dosing should follow the clinical effect. - start of preoxygenation with Bag-Valve-Mask Device or NIV when dissociative status is achieved for at least 3 minutes. - after completion of preoxygenation: neuromuscular blockade with Rocuronium - after application of Rocuronium: Intubation via standard of care. - should apnoea occur during preoxygenation, the continuation of ventilation via Bag-Valve-Mask or NIV is recommended, but not mandatory.
  Other Names: Delayed Sequence Intubation; DSI
  Arms: DSI
Procedure: Modified Rapid Sequence Induction — Modified Rapid Sequence Induction - Preoxygenation FiO2 100% with Bag-Valve-Mask-Device or NIV for at least 3 Minutes. - After completion of Preoxygeniation: application of Midazolam, Ketamin and Rocuronium. - The dosing of medication is determined in advance by the operating physician. - Ventilation via Bag-Valve-Mask-device or NIV after application of rocuronium is allowed. - After application of medication: Intubation via standard of care.
  Other Names: Rapid Sequence Intubation
  Arms: RSI

SUMMARY:
The goal of this clinical trial is to learn if it is feaseble to conduct a superiority trial comparing two methods for endotracheal intubation in critically ill patients. It will also learn about validity of outcomes regarding endotracheal intubation. The main questions it aims to answer are:

* Does performing intubation via Delayed Sequence Induction lower the incidence of severe hemodynamic complications compared to Rapid Sequence Induction?
* How are hemodynamic complications in the severely ill to be measured in order to minimize bias?

Participants will:

* receive emergency endotracheal intubation via Delayed or Rapid Sequence induction
* receive a phone call 90 days after endotracheal intubation
* outcome parameters outside of follow up phone calls will be routinely collected during the regular ICU-stay, there won't be any additional testing

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years or older in need of emergency endotracheal intubation in the following 60 minutes.
* The planned operateur routinely performs endotracheal intubation in critically ill patients.

Exclusion Criteria:

* Endotracheal Intubation performed during cardiopulmonary resuscitation or during "unstable ROSC", defined as Norepinephrine or Epinephrine dose > 0,5 µg/kgKG/min after return of spontaneous circulation.
* Participation in the study is not warranted because of increased risk for the patient or otherwise not justifiable (e.g. active oral bleeding).
* Known allergy against Ketamine, Esketamine, Midazolam or Rocuronium.
* Known contraindication against Ketamine, Esketamine Midazolam or Rocuronium.
* Known or anticipated difficult airway with indication for awake fiberoptic intubation.
* Women with known pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Collapse | From start of the procedure (= start of preoxygenation) until 60 minutes after start of the procedure.
  Composite Outcome:
  Hemodynamic Instability up to 60 minutes after start of the procedure, defined as:
  * any measured RRsyst < 65 mmHg or RRsyst < 90 mmHg for at least 30 minutes and/or
  * new need for Norepinephrine or increased dosage of Norepinephrine or need of a volume bolus > 15 ml/kgKG, to sustain a MAP > 65 mmHg/RR syst > 90 mmHg.
  and/or
  Cardiopulmonary Resuscitation up to 60 minutes after start of the procedure.

SECONDARY OUTCOMES:
Hemodynamic Instability | From start of the procedure (= start of preoxygenation) until 60 minutes after start of the procedure.
  Hemodynamic Instability up to 60 minutes after start of the procedure, defined as: - any measured RRsyst < 65 mmHg or RRsyst < 90 mmHg for at least 30 minutes and/or - new need for Norepinephrine or increased dosage of Norepinephrine or need of a volume bolus > 15 ml/kgKG, to sustain a MAP > 65 mmHg/RR syst > 90 mmHg.
Cardiopulmonary Resuscitation | From start of the procedure (= start of preoxygenation) until 60 minutes after start of the procedure.
  Cardiopulmonary Resuscitation, defined as any start of chest compressions.
spO2 after completion of preoxygenation | In both groups: spO2 at the time of application of rocuronium, which will be administered after preoxygenation has been completed and mark the beginning of the intubation procedure.
  spO2 [%] after completion of preoxygenation
Lowest spO2 during procedure | From start of the procedure (= start of preoxygenation) until confirmation of successful endotracheal intubation via waveform capnography or bronchoscopy, assessed up to 60 minutes.
  Lowest spO2 during procedure
Severe desaturation spO2 < 80% | From start of the procedure (= start of preoxygenation) until confirmation of successful endotracheal intubation via waveform capnography or bronchoscopy, assessed up to 60 minutes.
  Any spO2 measured below 80% during the intubation procedure.
Dose of Ketamine | From start of the procedure (= start of preoxygenation) until confirmation of successful endotracheal intubation via waveform capnography or bronchoscopy, assessed up to 60 minutes.
  Cumulative dose of Ketamine used.
Dose of Midazolam | From start of the procedure (= start of preoxygenation) until confirmation of successful endotracheal intubation via waveform capnography or bronchoscopy, assessed up to 60 minutes.
  Cumlative dose of Midazolam.
Endotracheal aspiration during intubation procedure | From start of the procedure (= start of preoxygenation) until confirmation of successful endotracheal intubation via waveform capnography or bronchoscopy, assessed up to 60 minutes.
  Endotracheal aspiration during intubation, defined as clinical observation by the intubating physician.
Number of intubation attempts | From start of the procedure (= start of preoxygenation) until confirmation of successful endotracheal intubation via waveform capnography or bronchoscopy, assessed up to 60 minutes.
  Cumulative number of intubation attempts. One attempt is defines as every new introduction of the laryngoskope through the open mouth.
New diagnosis of pneumonia | From start of the procedure (= start of preoxygenation) until 48 hours after start of the procedure.
  New diagnosis of pneumonia, defined as clinical interpretation of:
  * new infiltration in thoracic imaging (CT, chest xray, thoracic ultrasound)
  * proof of pathogen in respiratory material
  * worsening of oxygenation.
New diagnosis of pneumothorax | From start of the procedure (= start of preoxygenation) until 48 hours after start of the procedure.
  New diagnosis of pneumothorax, defined as:
  - proof of pneumothorax in thoracic imaging (CT, chest xray, thoracic ultrasound)
ICU-Mortality | From start of the procedure (= start of preoxygenation) until discharge from ICU, assessed up to 90 days.
  ICU-Mortality, defined as death during ICU-stay
Number of ICU-free days | From start of the procedure (= start of preoxygenation) until 90 days after start of the procedure.
  Number of days, in which the patient was alive outside any ICU.
Number of ventilator-free days | From start of the procedure (= start of preoxygenation) until 90 days after start of the procedure.
  Number of days, in which the patient was alive and free of invasive mechanical ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Anton J Pelka, Principal Investigator — Interdisciplinary Medical ICU, Leipzig Medical University Center
Locations (1):
- Interdisciplinary Medical ICU, Leipzig Medical University Center, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be allowed on reasonable request to the principal investigator after publication of the study results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be accessible after publication of the study results up to ten years.
Access Criteria: IPD will be accessible after obtaining the approval of the principal investigator on reasonable request. Access will be provided over a secured platform located at a LeipzigUMC server.